CLINICAL TRIAL: NCT01324752
Title: A Single-centre, Open-label, Three-period Study of the Pharmacokinetic Effect of PA21 on Losartan Potassium in Healthy Male and Female Adults
Brief Title: A Drug-Drug Interaction Study of Losartan and PA21
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PA-DDI-001
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Drug Interaction Potentiation
Keywords: Drug-drug interaction; Pharmacokinetics; PA21
MeSH Terms: interventions — Losartan; Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PA21 and Losartan with food (Experimental)
  Interventions: Drug: PA21 and Losartan with Food
- No PA21; Losartan with food (Experimental)
  Interventions: Drug: No PA21; Losartan with food
- PA21 with food and Losartan 2 hrs later (Experimental)
  Interventions: Drug: PA21 with food and Losartan 2 hours later

INTERVENTIONS:
Drug: PA21 and Losartan with Food — The maximum dose of PA21 will be 15.0 g/day. The maximum dose of Losartan will be 100 mg/day.
  Arms: PA21 and Losartan with food
Drug: No PA21; Losartan with food — The maximum dose of Losartan will be 100 mg/day.
  Arms: No PA21; Losartan with food
Drug: PA21 with food and Losartan 2 hours later — The maximum dose of PA21 will be 15.0 g/day. The maximum dose of Losartan will be 100 mg/day.
  Arms: PA21 with food and Losartan 2 hrs later

SUMMARY:
The purpose of this study is to determine if Losartan potassium is affected by PA21.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written informed consent

Exclusion Criteria:

* No significant medical conditions
* Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effect of PA21 on Losartan potassium | PK assessment on Day 0, 11, 22
  To assess the effect, if any, of PA21 on Losartan potassium exposure

SECONDARY OUTCOMES:
Effect of PA21 on the active metabolite of Losartan potassium | PK assessment on Day 0, 11, 22
  To assess the effect, if any, of PA21 on the active metabolite of Losartan potassium

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Winkle, MD, Principal Investigator — ACRI - Phase 1 (Advanced Clinical Research Institute)
Locations (1):
- ACRI- Phase 1, Anaheim, California, United States